CLINICAL TRIAL: NCT07245069
Title: Use of Dapagliflozin in Primary Prevention of Cardiotoxicity of Anthracycline Chemotherapy in Breast Cancer Patients
Acronym: Alpaca
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jure Tršan, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0120-383/2024-2711-3
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Anthracycline-induced Cardiac Toxicity; Endothelial Function (FMD); Arterial Stiffness; Breast Cancer
Keywords: Anthracycline-induced cardiac toxicity; Dapagliflozin; Breast Cancer; Cardio-Oncology; Primary Prevention; Global Longitudinal Strain; Myocardial Work; Endothelial Function; Flow-Mediated Dilation; Pulse Wave Velocity; Troponin; NT-proBNP; Heart Failure; Inflammation; Sodium-Glucose Transporter 2 Inhibitors
MeSH Terms: conditions — Heart Failure; Breast Neoplasms; Inflammation | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10 mg Daily (Experimental): Participants randomized to this arm will receive dapagliflozin 10 mg orally once daily for a total duration of 52 weeks (1 year). Study medication will begin before or at the start of anthracycline chemotherapy and will continue throughout chemotherapy and the post-treatment follow-up period, according to protocol.
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator): Participants randomized to this arm will receive a matching placebo orally once daily for a total duration of 52 weeks (1 year). Placebo will be initiated before or at the start of anthracycline chemotherapy and continued throughout chemotherapy and the 1-year protocol-defined follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Forgixa® 10 mg daily
  Arms: Dapagliflozin 10 mg Daily
Drug: Placebo — Lactose tablet daily
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to determine whether dapagliflozin, a sodium-glucose cotransporter-2 (SGLT-2) inhibitor, can help prevent anthracycline-induced cardiotoxicity caused by anthracycline chemotherapy in adult women with breast cancer receiving (neo)adjuvant treatment.

The main questions the study aims to answer are:

i) Does dapagliflozin reduce the decline in left ventricular function (measured by LVEF, GLS, and myocardial work) during and after anthracycline therapy? ii) Does dapagliflozin lessen the deteriorating effect of chemotherapy on endothelial function and arterial stiffness? iii) Does dapagliflozin effect levels of cardiac injury and inflammation biomarkers (e.g., hs-troponin T, NT-proBNP, ST-2, GDF-15, galectin-3, IL-6, MPO)?

Researchers will compare dapagliflozin 10 mg daily with placebo to see whether those receiving dapagliflozin experience less heart and vascular impairment during treatment.

Participants will:

* Take either dapagliflozin or placebo once daily during anthracycline chemotherapy.
* Undergo heart and vascular ultrasound, and a 6-minute walk test before chemotherapy and again at 24 and 52 weeks.
* Provide blood samples before, during and after chemotherapy to measure cardiac biomarkers.
* Complete multiple questionnaires on quality of life.

DETAILED DESCRIPTION:
Anthracycline-based chemotherapy remains a cornerstone of (neo)adjuvant treatment for breast cancer but is limited by a well-recognized risk of cardiotoxicity. This injury may manifest as left ventricular systolic dysfunction, abnormalities in myocardial deformation, impaired myocardial work efficiency, endothelial dysfunction, or increased arterial stiffness. Changes often occur early during treatment and may progress to clinically significant heart failure months or years after completion of chemotherapy. Current preventive strategies focus primarily on strict control of cardiovascular risk factors, as no pharmacologic intervention has consistently demonstrated efficacy in preventing anthracycline-induced cardiotoxicity.

SGLT-2 inhibitors, including dapagliflozin, have demonstrated robust cardiovascular benefits across diverse populations, independent of diabetes status. Clinical trials in heart failure and mechanistic studies indicate that SGLT-2 inhibition favorably affects myocardial energetics, reduces oxidative stress and inflammation, improves endothelial function, and modulates myocardial remodeling. Retrospective observational data in patients exposed to anthracyclines suggest fewer cardiac events among individuals using SGLT-2 inhibitors, but no prospective randomized trial has evaluated this potential cardioprotective effect.

This randomized, double-blind, placebo-controlled clinical trial is designed to determine whether dapagliflozin can attenuate cardiac and vascular deterioration associated with anthracycline chemotherapy in adults with breast cancer. Approximately 100 participants scheduled to receive four cycles of anthracycline-based (neo)adjuvant chemotherapy will be randomized (1:1) to receive dapagliflozin 10 mg once daily or matching placebo. Treatment will begin prior to or at the initiation of chemotherapy and continue according to protocol-defined duration.

Baseline evaluation includes transthoracic echocardiography with quantification of left ventricular ejection fraction (LVEF, using the modified biplane Simpson method), global longitudinal strain (GLS, via speckle-tracking in three apical views), and myocardial work indices derived from noninvasive blood pressure and strain analysis. Vascular ultrasonography will assess endothelial function through brachial artery flow-mediated dilation (FMD) and arterial stiffness via carotid pulse wave velocity (PWV) and stiffness index β. Functional capacity will be measured using the 6-minute walk test. Participants will also provide blood samples for a comprehensive biomarker panel including markers of myocardial injury (high-sensitivity troponin), hemodynamic stress (NT-proBNP), myocardial remodeling (ST-2, GDF-15, galectin-3), and inflammation (IL-6, myeloperoxidase). Quality of life will be assessed using EQ-5D, KCCQ, and SF-36 questionnaires.

All assessments (cardiac imaging, vascular studies, functional testing, and biomarker sampling) will be repeated at 24 and 52 weeks following initiation of chemotherapy, with an additional biomarker time point after two chemotherapy cycles and at the end of anthracycline treatment. This protocol enables characterization of both acute and subacute trajectories of myocardial and vascular injury.

The primary objective is to determine whether dapagliflozin reduces the degree of anthracycline-related left ventricular dysfunction, particularly reflected in GLS and myocardial work indices. Secondary objectives include evaluating effects on LVEF, endothelial function (FMD), arterial stiffness (PWV, stiffness β), biomarker profiles, functional capacity, and patient-reported outcomes. Safety monitoring will include systematic assessment of adverse events related to dapagliflozin, such as genitourinary infections, volume depletion, hypotension, and rare ketoacidosis. All participants will be monitored according to predefined stopping criteria and standard clinical safety procedures.

By integrating advanced cardiac and vascular phenotyping with serial biomarker profiling, this study aims to generate high-quality evidence on whether dapagliflozin provides meaningful primary prevention of anthracycline-induced cardiotoxicity. If beneficial, this approach could inform future cardio-oncology guidelines and improve cardiovascular safety for patients undergoing anthracycline chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Histologically confirmed breast cancer with planned (neo)adjuvant anthracycline-based chemotherapy (4 cycles of epirubicin + cyclophosphamide or doxorubicin + cyclophosphamide).
* Eligible to start dapagliflozin or placebo prior to or at initiation of chemotherapy.
* Able to perform baseline echocardiography, vascular ultrasound (FMD and carotid stiffness), 6-minute walk test, and biomarker sampling.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known heart failure (any prior diagnosis of HF).
* Clinically significant valvular heart disease.
* Prior exposure to chemotherapy or radiotherapy to the left chest.
* Type 1 diabetes mellitus.
* Symptomatic hypotension.
* History of recurrent urinary tract infections.
* History of diabetic ketoacidosis or ketonemia.
* Severe hepatic impairment (ALT, AST, ALP >3× upper limit of normal).
* Severe renal impairment (eGFR <20 mL/min/1.73 m²).
* Known allergy or intolerance to SGLT-2 inhibitors.
* Any use of SGLT-2 inhibitor therapy within 3 months prior to enrollment.
* Pregnancy or breastfeeding.
* Any condition that, in the investigator's judgment, could interfere with study participation, safety, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in Global Longitudinal Strain (GLS) | 52 weeks
  Global Longitudinal Strain (GLS), measured using speckle-tracking echocardiography in three apical views, will be used to quantify subclinical left ventricular systolic dysfunction. The primary endpoint is the change in GLS from baseline to 24 and 52 weeks. A relative worsening of >15% is considered clinically meaningful.
Change in Flow-Mediated Dilation (FMD) of the Brachial Artery | 52 weeks
  Endothelial function will be assessed by ultrasound measurement of flow-mediated dilation (FMD) of the brachial artery after forearm cuff occlusion. The endpoint is the absolute change in FMD (%) from baseline to 24 weeks. A reduction >2 absolute percentage points will be considered clinically meaningful. FMD will also be measured at 52 weeks to characterize the sustained effect of dapagliflozin on endothelial function compared with placebo.

SECONDARY OUTCOMES:
Change in Cardiovascular and Inflammatory Biomarkers | 52 weeks
  Serum concentrations of high-sensitivity cardiac troponin, NT-proBNP, ST-2, GDF-15, galectin-3, interleukin-6, and myeloperoxidase will be measured at predefined time points. The endpoint is the change in biomarker levels from baseline to 24 weeks, analyzed as absolute and/or relative change. Biomarkers will also be assessed at 52 weeks to evaluate longer-term effects of dapagliflozin on myocardial injury, hemodynamic stress, remodeling, and inflammation compared with placebo.
Change in Health-Related Quality of Life (EQ-5D Index Score) | 52 weeks
  Quality of life will be assessed using the EQ-5D questionnaire (5-dimension index score). The endpoint is the change in EQ-5D index score from baseline to 24 weeks. Higher scores indicate better health status. The questionnaire will also be administered at 52 weeks to evaluate longer-term effects of dapagliflozin versus placebo on patient-reported quality of life.
Change in Left Ventricular Ejection Fraction (LVEF) | 52 weeks
  LVEF will be measured by transthoracic echocardiography using the modified biplane Simpson method from apical 4- and 2-chamber views. The endpoint is the absolute change in LVEF (%) from baseline to 24 weeks. A decrease ≥10 percentage points or a drop below 53% will be considered clinically relevant. LVEF will also be assessed at 52 weeks to evaluate longer-term effects of dapagliflozin versus placebo on left ventricular systolic function.
Change in Carotid Arterial Stiffness (Pulse Wave Velocity and Stiffness Index β) | 52 weeks
  Arterial stiffness will be evaluated by ultrasound-based assessment of carotid pulse wave velocity (PWV) and stiffness index β using dedicated software. The endpoint is the absolute change in carotid PWV (m/s) and stiffness index β from baseline to 24 weeks. An increase in PWV ≥1 m/s will be considered clinically relevant. Measurements will be repeated at 52 weeks to assess persistent vascular effects of dapagliflozin versus placebo.
KCCQ (Kansas City Cardiomyopathy Questionnaire) | 52 weeks
  The KCCQ Overall Summary Score (0-100 scale) evaluates symptoms, physical limitations, social function, and quality of life related to cardiac health. The endpoint is the change in the Overall Summary Score from baseline to 24 weeks. A change ≥5 points is considered clinically meaningful. KCCQ will also be collected at 52 weeks to determine whether dapagliflozin influences patient-perceived cardiac function and symptom burden over time.
Change in SF-36 Health Survey Physical and Mental Component Summary Scores | 52 weeks
  Health-related quality of life will be evaluated using the SF-36 questionnaire, generating Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. The endpoint is the change in PCS and MCS from baseline to 24 weeks. Higher scores reflect better perceived health. SF-36 will also be administered at 52 weeks to assess sustained effects of dapagliflozin on global well-being and functional status.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia